CLINICAL TRIAL: NCT07006831
Title: A Multicenter, Prospective Blood Collection Study in a Kidney Transplant Population
Acronym: Accept cfDNA
Status: Recruiting | Type: Observational
Sponsor: Devyser Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DVYUS-TDX-001
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Kidney Disease; Kidney Transplant; Transplant Recipient; Renal Function; Cell-free DNA; NGS
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma from whole blood specimens and gDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: Kidney transplant recipients who are 18 years of age or older

SUMMARY:
The purpose of this research is to collect blood samples and data from kidney transplant patients. The samples and data will be used for research and development of non-invasive test to detect donor-derived cell-free DNA (dd-cfDNA) in kidney transplant patients to evaluate the status of the transplanted organ.

DETAILED DESCRIPTION:
This is a prospective, multicenter sample collection study within a kidney transplant population.

Whole blood samples and clinical data will be obtained from each participant at the time of indication biopsy (prior to the biopsy procedure).

De-identified leftover retrospective gDNA screening samples from the paired donor(s) will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Is 18 years of age or older at enrollment
3. Had a kidney transplant prior to enrollment
4. Is having an indication (for cause) biopsy as determined by clinician
5. retrospective leftover samples are available from the kidney donor(s).

Exclusion Criteria:

1. Is pregnant
2. Had a blood transfusion within the past 4 weeks
3. Had a transplant from an identical (monozygotic) twin
4. Had transplants of multiple organs from the same donor (eg, kidney and liver transplant).
5. Had transplants of more than 2 organs from different donors (eg, recipient of a third kidney transplant)
6. Had a transplant of hematopoietic stem cells (eg, bone marrow) or tissue (eg, heart valve)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Detection of donor-derived cell-free DNA (dd-cfDNA) from whole blood | 18 months
  Collected samples will be used for research and development of a noninvasive in- vitro diagnostic test to detect donor-derived cell-free DNA (dd-cfDNA) in kidney transplant patients.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Scripps Health, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Piedmont Healthcare, Atlanta, Georgia
  - University of Maryland Baltimore, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data with other researchers. Any shared data will be de-identified data at the cohort level in aggregate.

REFERENCES:
- [Background] Pettersson L, Westerling S, Talla V, Sendel A, Wennberg L, Olsson R, Hedrum A, Hauzenberger D. Development and performance of a next generation sequencing (NGS) assay for monitoring of dd-cfDNA post solid organ transplantation. Clin Chim Acta. 2024 Jan 1;552:117647. doi: 10.1016/j.cca.2023.117647. Epub 2023 Nov 10. PMID 37951377